CLINICAL TRIAL: NCT06303622
Title: A Randomised Controlled Trial Comparing MRI-Ultrasound Fusion and Cognitive-guided Biopsy for the Detection of Clinically Significant Prostate Cancer: the PROFUSION Trial
Brief Title: Comparing MRI-Ultrasound Fusion and Cognitive-guided Biopsy for the Detection of csPCa: the PROFUSION Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHIU Ka Fung Peter, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRE-2023.610
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRUS arm (Experimental): Targeted biopsies will be performed by software-assisted MRI-ultrasound fusion registration . Software-based fusion targeted biopsy of 4 cores per target followed by 12-core systematic biopsy will be performed. The fusion or overlay of 3D MRI and USG images create a detailed 3D prostate image with both targeted and systematic biopsy core locations recorded.
  Interventions: Procedure: MRI-USG fusion approach
- COG arm (Active Comparator): The biopsy operator reviews the MR images and creates a mental three-dimensional representation of the prostate and the lesion within it to guide biopsy. Cognitive registration is a visual guidance technique in which the surgeon samples a visually estimated location on transrectal ultrasound (TRUS) corresponding to the MRI suspicious regions. Cognitive-guided biopsy is performed by taking 4 cores from each target followed by 12-core systematic biopsies.
  Interventions: Procedure: Cognitive-guided approach

INTERVENTIONS:
Procedure: MRI-USG fusion approach — MRI-USG fusion approach prostate biopsy
  Arms: MRUS arm
Procedure: Cognitive-guided approach — Cognitive-guided approach prostate biopsy
  Arms: COG arm

SUMMARY:
This study is an international multicentre RCT to compare the linically significant prostate cancer (csPCa) detection of cognitive-guided and MRI-USG guided biopsies in men with suspicious MRI lesion.

DETAILED DESCRIPTION:
This study is an international multicentre RCT to compare the csPCa detection of cognitive-guided and MRI-USG guided biopsies in men with suspicious MRI lesion. This is a phase III randomised controlled trial to evaluate the detection of clinically significant prostate cancer (csPCa) by MRI-USG fusion approach (MRUS arm) versus Cognitive-guided approach (COG arm). The study hypothesis is that MRUS arm is superior to COG arm in detecting csPCa. The result of this RCT would impact how MRI-guided prostate biopsies should be done in the future. If the MRI-USG fusion approach is superior to cognitive-guidance in csPCa detection, it should be the standard of practice in the future, and dedicated MRI-USG fusion equipment should be available in centres performing prostate biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥18 years of age
* Clinical suspicion of prostate cancer and indicated for prostate biopsy
* Serum Prostate-specific antigen (PSA) < 20 ng/mL
* Digital rectal examination ≤ cT2 (organ-confined cancer)
* Able to provide written informed consent
* MRI prostate (contrast or plain) showing 1-3 suspicious lesion(s) with PI-RADS score 3-5

Exclusion Criteria:

* Prior prostate biopsy in the 2 years before screening visit
* Prior diagnosis of prostate cancer
* Contraindicated to prostate biopsy: active urinary tract infection, failed insertion of transrectal ultrasound probe into rectum (abdominal perineal resection, anal stenosis), uncorrectable coagulopathy, antiplatelet or anticoagulant which cannot be stopped (continue low-dose aspirin before and after biopsy is permitted)
* Patient refusal for biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 1250 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of men with clinically significant Prostate cancer(csPCa) | When histology results available, at an expected average of 30 days post-biopsy
  ISUP Grade 2 or above prostate cancer diagnosed on biopsy

SECONDARY OUTCOMES:
Proportion of men with a diagnosis of csPCa in MRI lesions with maximal size ≤10mm versus >10mm | When histology results available, at an expected average of 30 days post-biopsy
  MRI lesions with maximal size ≤10mm versus >10mm
Proportion of men with a diagnosis of csPCa in prostate size of ≤50ml vs >50m | When histology results available, at an expected average of 30 days post-biopsy
  prostate size of ≤50ml vs >50ml
The proportion of men with a diagnosis of csPCa only in targeted biopsy | When histology results available, at an expected average of 30 days post-biopsy
  ISUP Grade 2 or above prostate cancer diagnosed on biopsy
Proportion of men with a diagnosis of csPCa only in systemic biopsy | When histology results available, at an expected average of 30 days post-biopsy
  ISUP Grade 2 or above prostate cancer diagnosed on biopsy
Proportion of men with a diagnosis of clinically insignificant PCa, | When histology results available, at an expected average of 30 days post-biopsy
  ISUP grade group 1 Prostate cancer diagnosed on biopsy
Procedure time | During biopsy procedure
  Total time of procedure
Pain score on a scale of 0-10 taken after biopsy | Immediately After biopsy procedure
  The higher the score, the more pain
Proportion of men with post-biopsy adverse events within 30 days after biopsy | 30 days post biopsy
  The severity of Adverse event is grade by Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ka-Fungq CHIU, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Chan SY, Ng CF, Lee KW, Yee CH, Chiu PK, Teoh JY, Hou SS. Differences in cancer characteristics of Chinese patients with prostate cancer who present with different symptoms. Hong Kong Med J. 2017 Feb;23(1):6-12. doi: 10.12809/hkmj164875. Epub 2016 Dec 9. PMID 27932742
- [Background] Wong HF, Yee CH, Teoh JY, Chan SY, Chiu PK, Cheung HY, Hou SS, Ng CF. Time trend and characteristics of prostate cancer diagnosed in Hong Kong (China) in the past two decades. Asian J Androl. 2019 Jan 1;21(1):104-106. doi: 10.4103/aja.aja_75_18. No abstract available. PMID 30178778
- [Background] Patasius A, Smailyte G. Re: MaryBeth B. Culp, Isabelle Soerjomataram, Jason A. Efstathiou, Freddie Bray, Ahmedin Jemal. Recent Global Patterns in Prostate Cancer Incidence and Mortality Rates. Eur Urol 2020;77:38-52. Eur Urol. 2020 May;77(5):e132. doi: 10.1016/j.eururo.2019.11.030. Epub 2019 Dec 13. No abstract available. PMID 31843337
- [Background] Ahdoot M, Wilbur AR, Reese SE, Lebastchi AH, Mehralivand S, Gomella PT, Bloom J, Gurram S, Siddiqui M, Pinsky P, Parnes H, Linehan WM, Merino M, Choyke PL, Shih JH, Turkbey B, Wood BJ, Pinto PA. MRI-Targeted, Systematic, and Combined Biopsy for Prostate Cancer Diagnosis. N Engl J Med. 2020 Mar 5;382(10):917-928. doi: 10.1056/NEJMoa1910038. PMID 32130814
- [Background] Chiu PK, Alberts AR, Venderbos LDF, Bangma CH, Roobol MJ. Additional benefit of using a risk-based selection for prostate biopsy: an analysis of biopsy complications in the Rotterdam section of the European Randomized Study of Screening for Prostate Cancer. BJU Int. 2017 Sep;120(3):394-400. doi: 10.1111/bju.13913. Epub 2017 Jun 5. PMID 28498624
- [Background] Heidegger I, Pichler R. Re: Peter K.-F. Chiu, Chi-Fai Ng, Axel Semjonow, et al. A Multicentre Evaluation of the Role of the Prostate Health Index (PHI) in Regions with Differing Prevalence of Prostate Cancer: Adjustment of PHI Reference Ranges is Needed for European and Asian Settings. Eur Urol 2019;75:558-61. Eur Urol. 2019 Jun;75(6):e158-e159. doi: 10.1016/j.eururo.2018.12.041. Epub 2019 Jan 5. No abstract available. PMID 30616947
- [Background] Chiu PK, Roobol MJ, Nieboer D, Teoh JY, Yuen SK, Hou SM, Yiu MK, Ng CF. Adaptation and external validation of the European randomised study of screening for prostate cancer risk calculator for the Chinese population. Prostate Cancer Prostatic Dis. 2017 Mar;20(1):99-104. doi: 10.1038/pcan.2016.57. Epub 2016 Nov 29. PMID 27897172
- [Background] Turkbey B, Rosenkrantz AB, Haider MA, Padhani AR, Villeirs G, Macura KJ, Tempany CM, Choyke PL, Cornud F, Margolis DJ, Thoeny HC, Verma S, Barentsz J, Weinreb JC. Prostate Imaging Reporting and Data System Version 2.1: 2019 Update of Prostate Imaging Reporting and Data System Version 2. Eur Urol. 2019 Sep;76(3):340-351. doi: 10.1016/j.eururo.2019.02.033. Epub 2019 Mar 18. PMID 30898406
- [Background] Alberts AR, Roobol MJ, Verbeek JFM, Schoots IG, Chiu PK, Osses DF, Tijsterman JD, Beerlage HP, Mannaerts CK, Schimmoller L, Albers P, Arsov C. Prediction of High-grade Prostate Cancer Following Multiparametric Magnetic Resonance Imaging: Improving the Rotterdam European Randomized Study of Screening for Prostate Cancer Risk Calculators. Eur Urol. 2019 Feb;75(2):310-318. doi: 10.1016/j.eururo.2018.07.031. Epub 2018 Aug 3. PMID 30082150
- [Background] Drost FH, Osses DF, Nieboer D, Steyerberg EW, Bangma CH, Roobol MJ, Schoots IG. Prostate MRI, with or without MRI-targeted biopsy, and systematic biopsy for detecting prostate cancer. Cochrane Database Syst Rev. 2019 Apr 25;4(4):CD012663. doi: 10.1002/14651858.CD012663.pub2. PMID 31022301
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975
- [Background] Connor MJ, Gorin MA, Eldred-Evans D, Bass EJ, Desai A, Dudderidge T, Winkler M, Ahmed HU. Landmarks in the evolution of prostate biopsy. Nat Rev Urol. 2023 Apr;20(4):241-258. doi: 10.1038/s41585-022-00684-0. Epub 2023 Jan 18. PMID 36653670
- [Background] Chiu PK, Roobol MJ, Teoh JY, Lee WM, Yip SY, Hou SM, Bangma CH, Ng CF. Prostate health index (PHI) and prostate-specific antigen (PSA) predictive models for prostate cancer in the Chinese population and the role of digital rectal examination-estimated prostate volume. Int Urol Nephrol. 2016 Oct;48(10):1631-7. doi: 10.1007/s11255-016-1350-8. Epub 2016 Jun 27. PMID 27349564
- [Background] Gigot O. [Treatment of alcoholic intoxication (exclusive of acute attacks)]. Infirm Fr. 1970 Jun;116:31 passimc. No abstract available. French. PMID 5201460
- See also: Hong Kong Cancer Statistics — https://www3.ha.org.hk/cancereg/pdf/factsheet/2019/prostate_.pdf